CLINICAL TRIAL: NCT06745180
Title: Making Healthy Habits Stick: Extended Contact Interventions to Promote Long-Term Physical Activity in Cancer Survivors
Brief Title: Making Healthy Habits Stick
Acronym: HABITS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB-300011855; R01MD018375 (NIH)
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Physical Activity; Cancer Survivor; Cancer Survivorship
Keywords: Physical Activity; Cancer; Cancer Survivor; Exercise; Cancer Survivorship
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Spermine Synthase

STUDY DESIGN:
Intervention Model Description: 2x2 Factorial Design
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Peer Coach and SMS (Experimental): SMS and peer coach interventions focused on physical activity maintenance
  Interventions: Behavioral: Peer Coach and SMS
- Peer Coach (Experimental): Peer coach intervention focused on physical activity maintenance
  Interventions: Behavioral: Peer Coach
- Short Message Service (SMS) (Experimental): SMS intervention focused on physical activity maintenance
  Interventions: Behavioral: Short Message System (SMS)
- Usual Care (Other): Written materials focused on physical activity maintenance
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Short Message System (SMS) — The Short Message System (SMS) intervention focuses on personalized, adaptive SMS messages that help the participant maintain physical activity behaviors.
  Other Names: SMS; Short Message Service
  Arms: Short Message Service (SMS)
Behavioral: Peer Coach — The peer coach will deliver an intervention that will help participants maintain physical activity.
  Other Names: Peer Support; Peer Sustainability
  Arms: Peer Coach
Behavioral: Usual Care — Participants will be given written materials providing advice on maintaining their physical activity.
  Arms: Usual Care
Behavioral: Peer Coach and SMS — The Short Message System (SMS) intervention focuses on personalized, adaptive SMS messages that help the participant maintain physical activity behaviors. The peer coach will deliver an intervention that will help participants maintain physical activity.
  Arms: Peer Coach and SMS

SUMMARY:
The aim of this project is to help increase physical activity maintenance in cancer survivors.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate novel interventions designed to assist women cancer survivors, who identify as African American or Black, in overcoming exercise barriers, developing a physically active mindset, and establishing exercise habits needed to exercise long term. These novel interventions are 1. Text Messaging (SMS), 2. Peer Coaching, 3. Combination of Peer Coaching and SMS, 4. Usual Care

ELIGIBILITY:
Inclusion Criteria:

* woman age of 19 or older
* identifies as African American or Black
* have a history of cancer
* have completed post-primary treatment for cancer (i.e., chemotherapy, radiation)
* agree to allow research team to confirm cancer diagnosis with your physician
* If received surgery, must be at least 8 weeks post-surgery
* willing to have regular physician provide medical clearance for study participation
* willing to provide home address if qualified for the study
* willing and able to use videoconference platform such as Zoom for study activities (must be both willing and able)
* willing and able to send and/or receive text messages (must be both willing and able)
* has US phone number
* has an email address
* if has no email address, must be willing to create one
* English speaking
* Able to ambulate without assistance (does not need to use a cane, a walker, or a wheelchair)
* willing and able to complete 3-5 exercise session per week on their own for the duration of the study; if answered no, please explain
* willing to attend individual and group sessions via videoconferences during study participation; if answered no, please explain.
* willing to attend assessments via videoconference during study participation; if answered no, please explain.
* willing to complete surveys during study participation; if answered no, please explain.

Exclusion Criteria:

* Metastatic or recurrent cancer
* another cancer diagnosis in the past 5 years (not including skin or cervical cancer in situ)
* have severe orthopedic, joints or any other condition that stops individual from being active
* unstable angina
* have paint, tightness, or heaviness in chest EITHER when resting OR then physically active
* have New York Heart Association class II, III, OR IV congestive heart failure
* blood pressure has been over 160/100 at least twice in the past 6 months (either number; 160 or 100)
* have uncontrolled asthma
* have interstitial lung disease that requires extra oxygen
* have dementia or organize brain syndrome
* have schizophrenia or active psychosis
* have had a stroke or other problem that left individual disables or with paralysis (unable to move or feel any part of body)
* have hearing problems that make it hard to carry on a phone conversation
* blind or partially blind
* planned surgery during the first 6 month of study participation (if unapproved by PI)
* planned knee or hip surgery during the first 6 month of study participation
* anticipate changes in usual medications during the first 6 months of study participation (if unapproved by PI)
* have been told by a physician to only do exercise prescribed by a physician
* have been told by a physician to limit physical activity
* have a contraindication to engaging in moderate intensity aerobic exercise
* have completed on average, more than 90 min/week of moderate-intensity or more that 30 min/week of vigorous exercise in the past 6 months
* trouble with balance or moving around safely
* are currently pregnant or anticipate pregnant during study participation
* currently participating in another exercise study
* have BMI ≥ 50

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Physical Activity (patient reported outcome) | From Baseline to 15 Month Assessment
  Participants will wear motion sensor on waist for 7 days

SECONDARY OUTCOMES:
Fatigue (Patient reported outcome) | At Baseline, 3 month assessment, 9 month assessment, and 15 month assessment.
  Fatigue will be measured using the Fatigue Symptom Inventory (fatigue intensity and interference) scale.
Self-perceived Health (Patient reported outcome) | At Baseline, 3 month assessment, 9 month assessment, and 15 month assessment.
  Self-perceived health will be measured using the EQ-5D questionnaire.
Qualify of life (Patient reported outcome) | At Baseline, 3 month assessment, 9 month assessment, and 15 month assessment.
  Quality of life will be measured via the PROMIS Global Health questionnaire.
Anxiety & Depression (patient reported outcome) | At Baseline, 3 month assessment, 9 month assessment, and 15 month assessment.
  Anxiety and depression will be measured using the Hospital Anxiety and Depression Scale.

OTHER OUTCOMES:
Stress (patient reported outcome) | At Baseline, 3 months, 9 months, and 15 months
  Stress will be measured using the Perceived Stress Scale
Social Determinants of Health | At Baseline, 3 months, 9 months, 15 months
  Social determinants of health will be measured using the Social Determinants of Health (SDoH) questionnaire.
Big Five Personality (patient reported outcome) | At Baseline, 3 months, 9 months, 15 months
  Big five personality will be measured using a brief version of the Big Five Personality Inventory questionnaire.
Self-report Physical Activity | At Baseline, 3 months, 9 months, 15 months
  Aerobic and resistance exercise will be measured using the Godin Aerobic Strength questionnaire.
Quality of Life (patient reported outcome) | At Baseline, 3 months, 9 months, 15 months
  Quality of life will be measured using the EQ-5D-5L questionnaire.
Social Support for Physical Activity (patient reported outcome) | At Baseline, 3 months, 9 months, 15 months
  Social support for physical activity will be measured using the Social Support for PA questionnaire.
Reflective, Regulatory, and Reflexive processes (patient reported outcome) | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months
  Reflective, regulatory, and reflexive processes is being measured by the M-PAC physical activity questionnaire.
Perceived Exercise Barriers Interference | At Baseline, 3 months, 9 months, 15 months
  Barriers to exercise will be measured using the Perceived Barriers to Exercise questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Martin, PhD, Principal Investigator — University of Tennessee; Laura Rogers, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Tennessee Health Science Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individuals interested in requesting IPD should contact the study PIs.
Supporting Information: ICF
Time Frame: After data management is finalized (and data locked) and the manuscript reporting physical activity maintenance data at month 15 has been submitted
Access Criteria: A data use agreement between the institution housing the data (UTHSC) and the institution of the requesting researcher will be required.

DOCUMENTS (1):
  • Study Protocol (2024-11-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT06745180/Prot_000.pdf